CLINICAL TRIAL: NCT04793243
Title: Vitamin D3 Levels in COVID-19 Outpatients From Western Mexico: Clinical Correlation and Effect of Its Supplementation
Brief Title: Vitamin D3 Levels in COVID-19 Outpatients From Western Mexico
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Jose Francisco Munoz Valle, Provost of the University Center of Health Sciences, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CI-07620
Record Dates: First submitted 2021-03-03; First posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Covid19
Keywords: vitamin D; Latin America; supplementation
MeSH Terms: conditions — COVID-19 | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Formed by 22 patients that received oral supplementation of 10,000 IU daily for fourteen days of vitamin D3
  Interventions: Dietary Supplement: Vitamin D3
- Control group (No Intervention): Formed by 20 patients that did not receive supplementation

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Patients received oral supplementation of 10,000 IU daily for fourteen days of vitamin D3
  Arms: Intervention group

SUMMARY:
The immunomodulatory effects of vitamin D are known to be beneficial in viral infections, it is also known that its deficiency is associated with a worse prognosis of COVID-19. This study aimed to determine the baseline vitamin D serum concentrations in asymptomatic or mildly symptomatic COVID-19 outpatients, as well as to evaluate the effects of supplementation with 10,00 IU/daily of vitamin D3 and its relationship with biochemical parameters and clinical features.

ELIGIBILITY:
Inclusion criteria:

* Intervention group: Patients with positive PCR for COVID-19 of both sexes supplemented with vitamin D
* Control group: Patients with positive PCR for COVID-19 of both sexes
* Both groups: Mexican individuals, after signing the informed consent letter and over 18 years of age.

Exclusion criteria:

• Diseases that compromise the absorption of Vitamin D; Crohn's disease, cystic fibrosis, and celiac disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2020-10-10 (Actual); Study Completion 2020-10-24 (Actual)

PRIMARY OUTCOMES:
Baseline levels of serum vitamin D in COVID-19 patients | At baseline
  Evaluate serum levels of 25(OH)D (ng/mL) in patients with covid-19 from western Mexico
Correlation between D-dimer and vitamin D serum levels in COVID-19 patients | At baseline
  Serum levels of D-dimer (ng/mL) will be measured at baseline and correlated with levels of 25(OH)D (ng/mL) in patients with covid-19 from western Mexico
Correlation between transferrin and vitamin D serum levels in COVID-19 patients | At baseline
  Serum levels of transferrin (mg/dL) will be measured at baseline and correlated with levels of 25(OH)D (ng/mL) in patients with covid-19 from western Mexico
Correlation between ferritin and vitamin D serum levels in COVID-19 patients | At baseline
  Serum levels of ferritin (ng/mL) will be measured at baseline and correlated with levels of 25(OH)D (ng/mL) in patients with covid-19 from western Mexico
Effects of vitamin D3 supplementation on COVID-19 patients | After 14 days of supplementation
  Serum levels of 25(OH)D (ng/mL) will be determined in the intervention group after 14 days of Vitamin D3 supplementation

CONTACTS AND LOCATIONS:
Overall Officials: José F Muñoz-Valle, Dr., Principal Investigator — University of Guadalajara
Locations (1):
- Universidad de Guadalajara, Guadalajara, Jalisco, Mexico